CLINICAL TRIAL: NCT05859048
Title: Multidisciplinary Approach for High Risk Patients Leading to Early Diagnosis of Canadians
Brief Title: Multidisciplinary Approach for High Risk Patients Leading to Early Diagnosis of Canadians in Heart Failure
Acronym: MAPLE-CHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiology Research UBC (Other)
Collaborators: AstraZeneca (Industry); Centre for Cardiovascular Innovation (Unknown); NHS Greater Glasgow & Clyde (Unknown); HeartLife Foundation (Unknown); Canadian Heart Function Alliance (Unknown); Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Nathaniel Hawkins, Principal Investigator, Cardiology Research UBC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MAPLE-CHF
Record Dates: First submitted 2023-05-01; First posted 2023-05-15 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
Keywords: Heart failure screening; natriuretic peptides; artificial intelligence echocardiography
MeSH Terms: conditions — Heart Failure | interventions — Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational arm guided by NT-proBNP result (Active Comparator): NT-proBNP drawn and if level elevated (>125 pg/ml) a study visit with artificial intelligence (AI) echocardiogram, electrocardiogram (ECG), and heart failure (HF) focused examination conducted
  Interventions: Diagnostic Test: NT-proBNP; Diagnostic Test: AI echocardiogram; Diagnostic Test: electrocardiogram; Other: Cardiovascular physical examination
- Routine care arm (No Intervention): Participants will be remotely monitored for number of heart failure events

INTERVENTIONS:
Diagnostic Test: NT-proBNP — blood sample to measure N-terminal prohormone of B-type natriuretic peptide at local laboratory
  Arms: Investigational arm guided by NT-proBNP result
Diagnostic Test: AI echocardiogram — Artificial intelligence driven transthoracic echocardiogram
  Arms: Investigational arm guided by NT-proBNP result
Diagnostic Test: electrocardiogram — tracing of electrical cardiac activity of the heart
  Arms: Investigational arm guided by NT-proBNP result
Other: Cardiovascular physical examination — basic physiological measurements to include height (cm), weight (kg) and hip circumference (cm) and blood pressure (mmHg)
  Arms: Investigational arm guided by NT-proBNP result

SUMMARY:
The goal of this study is improve the screening of heart failure and identify patients early who are at risk of heart failure.

The main question[s] it aims to answer are:

• will an electronic health records (EHR) case finding algorithm for heart failure, followed by N-Terminal pro-brain natriuretic peptide (NT-proBNP) screening and artificial intelligence (AI) echocardiogram compared to usual care identify patients at risk for heart failure earlier than standard of care?

Participants will be enrolled and randomized to either standard of care (SOC) or intervention arm:

SOC arm: electronic health records will be reviewed over six months for assessments performed to identify heart failure.

Intervention arm: blood sample for N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) at local laboratory . For elevated NT-proBNP results (>125pg/ml) an artificial intelligence (AI) echocardiogram and 12 lead electrocardiogram (ECG) will be performed at study site (within 28 days of NT-proBNP result). EHR will be reviewed at six months

DETAILED DESCRIPTION:
Heart failure describes a chronic condition where the heart muscle is no longer able to supply the body with enough oxygen and nutrients. This can lead to fatigue and poor quality of life. Often, people do not know they have heart failure until they end up in hospital. This study wants to improve the screening of heart failure and identify patients at risk for heart failure earlier. This will help determine if early-screening and treatment can help prevent further decline in these patients.

This is a randomized, un-blinded study comparing usual care to an intervention group receiving early heart failure testing. Pre-screening will be performed using extracted primary care electronic health records with the case finding algorithm based on the inclusion and exclusion criteria. An invitation letter will be send to prospective patients which include a registration telephone number and link to dedicated study website. The invitation for contact will adopt an "opt out" approach (ask the potential participant to contact the coordinating centre if they do not wish to be contacted).

Potential participants not opting out, or opting in, within 2 weeks of invitation mailing will be sent a patient information package along with follow up contact by research team.

Consented participants will be randomized either to usual care or interventions group and followed for six months. Intervention group will have NT-proBNP drawn and those with an elevated NT-proBNP (>125pg/mL) will have a study visit with assessments to include, physical examination, electrocardiogram and study AI echocardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 40 years of age
* Informed consent
* At least two additional risk factors for Heart Failure (HF):

  * Coronary artery disease (either a previous documented type 1 myocardial infarction or coronary artery bypass grafting or percutaneous coronary intervention or documented stenosis or an epicardial coronary artery (50% left main stem or >70% left anterior descending, circumflex or right coronary artery)).
  * Diabetes type 1 or 2.
  * Persistent or permanent atrial fibrillation.
  * Previous ischemic or embolic stroke.
  * Peripheral artery disease (previous surgical or percutaneous revascularization or documented stenosis >50% of major peripheral arterial vessel.
  * Chronic kidney disease (defined as an estimated glomerular filtration rate (eGFR)<60 milliliters per minute (mL/min)/1.73m2 or eGFR 60-90 mL/min/1.73m2 and urine albumin-creatinine ration (UACR) >300mg/g).
  * Regular loop diuretic use for >30 days within 12 months prior to consent.
  * Chronic obstructive pulmonary disease (COPD) evidenced by one of the following: Pulmonary Function Test (PFT) showing airway obstruction, diagnosis of respiratory physician, CT scan reporting presence of emphysema, or treatment with national guidance advocated COPD therapy.

Exclusion Criteria:

* Inability to give informed consent (e.g. due to significant cognitive impairment).
* Previous diagnosis of heart failure. This is any diagnosis of heart failure with any ejection fraction of any cause.
* Renal replacement therapy.
* Anyone who, in the investigator's opinion, is not suitable to participate in the trial for other reasons e.g., a diagnosis which may compromise survival over the study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1360 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants diagnosed with heart failure (HF) according to the European Society of Cardiology 2021 HF guidelines | enrollment to six months
  Incidence of HF diagnosis in outpatient settings Urgent heart failure visit. Heart failure hospitalization.
Number of outpatient HF visits | enrollment to six months
  Number of outpatient visits for HF with initiation or intensification of oral HF therapy
Number of urgent HF visit | enrollment to six months
  Incidence of HF presentation in urgent care setting with administration of intravenous HF therapies
Number of HF hospitalizations | enrollment to six months
  Number of admission for HF

SECONDARY OUTCOMES:
incidence of prescription for guideline recommended HF therapies in patients diagnosed with HFrEF | enrollment to six months
  number of diagnosis of HF with reduced Ejection Fraction (HFrEF) within 6 months.
  Patients diagnosed with HFrEF receiving Guideline-directed medical therapy within 6 months
HF events in HFrEF | enrollment to six months
  number of HF admissions

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel M Hawkins, MD, Principal Investigator — Associate Professor of Medicine, UBC Division of Cardiology; Anique Ducharme, MD, Principal Investigator — Professor of Medicine, Univeriste de Montreal, Montreal Heart Institute; Serge LePage, MD, Principal Investigator — Centre Hospitalier Universite de Sherbrooke-Hopital Fleurimont
Locations (3):
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Montreal Heart Institute, Montreal, Quebec
  - University of Sherbrooke, Sherbrooke, Quebec